CLINICAL TRIAL: NCT03160703
Title: A Proof of Principal Study to Investigate the Stain Control of Two Stannous Fluoride Dentifrices
Brief Title: Study to Investigate the Stain Control of Two Stannous Fluoride Dentifrices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 207872
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Results first posted 2019-01-17 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Extrinsic Dental Stain; Oral Hygiene
Keywords: Dental stain, stannous fluoride, dentifrice
MeSH Terms: interventions — Tin Fluorides; triphosphoric acid; fluorophosphate

STUDY DESIGN:
Intervention Model Description: Single centre, randomised, examiner blind, parallel design study to evaluate the buildup of extrinsic dental stain over a 4 week treatment period
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test dentifrice 1 (RDA~58) (Experimental): Participants will apply experimental dentifrice containing 0.454% SnF2 / 5% STP.
  Interventions: Other: Stannous fluoride (SnF2, 0.454%), Sodium tripolyphosphate (STP, 5%), 2.0% abrasive silica
- Test dentifrice 2 (RDA~77) (Experimental): Participants will apply experimental dentifrice containing 0.454% SnF2 / 5% STP.
  Interventions: Other: Stannous fluoride (SnF2, 0.454%), Sodium tripolyphosphate (STP, 5%), abrasive silica (3.5%)
- Reference dentifrice 1 (RDA~80) (Other): Participants will apply dentifrice containing 1000 parts per million (ppm) fluoride as Sodium Monofluorophosphate (SMFP).
  Interventions: Other: Sodium Monofluorophosphate (1000 ppm fluoride ), RDA~80
- Reference dentifrice 2 (RDA~120) (Active Comparator): Participants will apply dentifrice containing 0.454% SnF2.
  Interventions: Other: Stannous fluoride (SnF2, 0.454%), RDA~120

INTERVENTIONS:
Other: Stannous fluoride (SnF2, 0.454%), Sodium tripolyphosphate (STP, 5%), 2.0% abrasive silica — Participants will apply a full brush head of their dentifrice containing 0.454% SnF2 / 5% STP; 2.0% abrasive silica (RDA~58) and will brush twice daily (morning and evening) for one timed minute (in their usual manner) and expectorate.
  Arms: Test dentifrice 1 (RDA~58)
Other: Stannous fluoride (SnF2, 0.454%), Sodium tripolyphosphate (STP, 5%), abrasive silica (3.5%) — Participants will apply a full brush head of their dentifrice containing 0.454% SnF2 / 5% STP; 3.5% abrasive silica (RDA~77) and will brush twice daily (morning and evening) for one timed minute (in their usual manner) and expectorate.
  Arms: Test dentifrice 2 (RDA~77)
Other: Sodium Monofluorophosphate (1000 ppm fluoride ), RDA~80 — Participants will apply a full brush head of their dentifrice containing 1000 ppm fluoride as SMFP with moderate abrasivity (RDA~80) and will brush twice daily (morning and evening) for one timed minute (in their usual manner) and expectorate.
  Arms: Reference dentifrice 1 (RDA~80)
Other: Stannous fluoride (SnF2, 0.454%), RDA~120 — Participants will apply a full brush head of their dentifrice containing 0.454% SnF2 with higher abrasivity (RDA~120) and will brush twice daily (morning and evening) for one timed minute (in their usual manner) and expectorate.
  Arms: Reference dentifrice 2 (RDA~120)

SUMMARY:
The purpose of this study is to evaluate and compare the stain build up of two stannous fluoride (SnF2) / sodium tripolyphosphate (STP) dentifrices of differing abrasivity levels, with a marketed standard fluoride dentifrice and a marketed SnF2 dentifrice.

DETAILED DESCRIPTION:
This proof of principal (PoP) single centre, randomised, examiner blind, four-treatment arm, parallel design study will be used to evaluate and compare the stain buildup of two 0.454% SnF2/ 5% STP dentifrices of differing abrasivity levels, with a marketed standard fluoride dentifrice and a marketed SnF2 dentifrice. Stain will be assessed following a full professional dental prophylaxis, at intervals over a 4 week treatment period, using an established clinical measure of extrinsic dental stain - the MacPherson modification of the Lobene stain index (MLSI). Participants will be stratified by pre-prophylaxis MLSI score (total MLSI Area x Intensity (A×I) for the facial surfaces of the 12 anterior teeth) and smoking status. The study will be conducted in healthy participants with a propensity for extrinsic dental stain (in the opinion of the examiner) on the facial surfaces of the anterior teeth.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Understands and is willing, able and likely to comply with all study procedures and restrictions.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee: No clinically significant and relevant abnormalities of medical history or oral examination which could impact study outcomes, Absence of any condition that would impact on subject safety or wellbeing, or affect the subject's ability to understand and follow study procedures and requirements.
* In the opinion of the investigator or medically qualified designee, At screening: Good oral health, at least 16 natural teeth including the 12 anterior teeth, the facial surfaces, and mandibular lingual surfaces, of at least 11 of the 12 anterior teeth, gradable for the MLSI, presence of extrinsic dental stain (judged to be formed due to dietary factors, or use of tobacco products) on the facial surfaces of the anterior teeth, as determined from a visual stain assessment. At baseline: A sufficient level of extrinsic dental stain (in the opinion of the examiner) on the facial surfaces of the scorable anterior (maxillary and mandibular) teeth.

Exclusion Criteria:

* Women who are known to be pregnant, or who are intending to become pregnant over the duration of the study. Since this study is not being conducted under an IND this information will be self-reported, and not diagnosed through the conduct of urinary pregnancy testing.
* Women who are breast-feeding.
* Recent history (within the last year) of alcohol or other substance abuse.
* Concurrent Medication: Current regular use of mouthwashes containing ingredients that are known to impart staining. For example, chlorhexidine or cetylpyridinium chloride (CPC), Use of minocycline, tetracycline or doxycycline within 30 days prior to screening, Use of minocycline, tetracycline or doxycycline between the screening and baseline visit, Daily doses of a medication and/or traditional/herbal ingredients which, in the opinion of the investigator, may affect study outcomes. For example, drugs or supplements containing metal ions known to impart staining to the enamel.
* Disease: Presence of chronic debilitating disease which, in the opinion of the investigator, could affect study outcomes, Any condition which, in the opinion of the investigator, causes xerostomia.
* Allergy/Intolerance:Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Clinical study/Experimental Product:Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit, Previous participation in this study.
* General dentition exclusions: Dental prophylaxis within 8 weeks of screening, Gross periodontal disease, treatment of periodontal disease (including surgery) within 12 months of screening, scaling or root planning within 3 months of screening, Use of any professionally dispensed or over the counter bleaching/ whitening products (excluding daily use whitening dentifrices) within the past 3 months.
* Specific Dentition Exclusions for Test Teeth: Any tooth which, in the opinion of the investigator, appears to be non-vital based on changes in the intrinsic colour, tooth with evidence of current or recent caries, or reported treatment of decay in 12 months of screening, tooth with exposed dentine which, in the opinion of the investigator, could impact grading of extrinsic dental stain; tooth with deep, defective or facial restorations; tooth used as an abutment for fixed or removable partial dentures; tooth with full crown or veneer, orthodontic bands or cracked enamel, tooth with surface irregularities, discoloration due to trauma, tetracycline stain, restorations, or hypo or hyperplasic areas which, in the opinion of the investigator, would prevent consistent grading of extrinsic dental stain.
* Personnel: An employee of the sponsor or the study site or members of their immediate family.
* Other: Any subject who, in the judgment of the investigator, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mason S, Young S, Qaqish J, Frappin G, Goyal C. Stain control with two modified stannous fluoride/sodium tripolyphosphate toothpastes: A randomised controlled proof of concept study. J Dent. 2019;91S:100009. doi: 10.1016/j.jjodo.2019.100009. Epub 2019 Oct 7. PMID 34059275

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one center in Canada.
Pre-assignment Details: A total of 225 participants were screened, of which 220 participants were enrolled and randomized in the study. A total of 5 participants were not randomized in study as 3 participants did not meet study criteria, and 2 withdrew their consent.
Groups:
- Test Dentifrice 1 (RDA~58): Participants applied experimental dentifrice containing 0.454 percent (%) stannous fluoride (SnF2) / 5% sodium tripolyphosphate (STP); 2.0% abrasive silica
- Test Dentifrice 2 (RDA~77): Participants applied experimental dentifrice containing 0.454% SnF2 / 5% STP; 3.5% abrasive silica
- Reference Dentifrice 1 (RDA~80): Participants applied dentifrice containing 1000 parts per million (ppm) fluoride as Sodium Monofluorophosphate (SMFP)
- Reference Dentifrice 2 (RDA~120): Participants applied dentifrice containing 0.454% SnF2
Period: Overall Study
Arm/Group | Test Dentifrice 1 (RDA~58) | Test Dentifrice 2 (RDA~77) | Reference Dentifrice 1 (RDA~80) | Reference Dentifrice 2 (RDA~120)
Started | 55 | 55 | 55 | 55
Completed | 55 | 55 | 55 | 54
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Test Dentifrice 1 (RDA~58): Participants applied experimental dentifrice containing 0.454% SnF2 / 5% STP; 2.0% abrasive silica
- Reference Dentifrice 1 (RDA~80): Participants applied dentifrice containing 1000 ppm fluoride as SMFP
- Total: Total of all reporting groups
Arm/Group | Test Dentifrice 1 (RDA~58) | Test Dentifrice 2 (RDA~77) | Reference Dentifrice 1 (RDA~80) | Reference Dentifrice 2 (RDA~120) | Total
Number analyzed (Participants) | 55 | 55 | 55 | 55 | 220
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.3 (10.80) | 46.1 (11.20) | 48.7 (11.50) | 46.6 (12.28) | 47.7 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 39 | 40 | 44 | 159
  Male | 19 | 16 | 15 | 11 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 12 | 13 | 11 | 5 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 20 | 17 | 10 | 15 | 62
  White | 23 | 24 | 33 | 35 | 115
  More than one race | 0 | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Modified Lobene Stain Index (MLSI) Mean Score at Week 4
Description: An assessment of the area and intensity of dental stain on the study teeth was performed using the MLSI after usage of the allocated study dentifrice, after 4 weeks twice daily use. The intensity of stain was scored separately for the gingival and body areas of each assessable tooth on a scale of 0 to 3 (0 - no stain, 1- light stain, 2 - moderate stain, 3 - heavy stain). The area of stain was scored separately for the gingival and body areas of each assessable tooth on the following scale: 0 - no stain; 1 - stain up to 1/3 of the area affected; 2- stain between 1/3 and 2/3 of the area affected; and 3 - stain more than 2/3 of area affected. Overall MLSI was calculated by multiplying scores of intensity and area, and was thus analyzed on a scale of 0 (best score) to 9 (worst score).
Time Frame: Baseline and Week 4
Population: The Intent-To-Treat (ITT) population (N=219) included all participants who were randomized, received at least 1 dose of investigational product, and had at least 1 post-baseline efficacy evaluation and were reported by randomized treatment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Test Dentifrice 1 (RDA~58) | Test Dentifrice 2 (RDA~77) | Reference Dentifrice 1 (RDA~80) | Reference Dentifrice 2 (RDA~120)
Number analyzed (Participants) | 55 | 55 | 55 | 54
Score on a scale
  Baseline | 1.38 (0.423) | 1.43 (0.422) | 1.42 (0.626) | 1.38 (0.443)
  Week 4 | 0.08 (0.078) | 0.05 (0.057) | 0.10 (0.096) | 0.16 (0.141)
Statistical Analysis 1: Comparison: Test Dentifrice 1 (RDA~58) vs Reference Dentifrice 1 (RDA~80); Test type: Superiority; p = 0.2681, ANCOVA — Statistical significance set at 5% level; From ANCOVA with treatment and smoking status as factors and baseline pre-prophylaxis overall MLSI score as covariate; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.05 to 0.01] — Difference is first named treatment minus second named treatment such that a negative difference favours the first named treatment
Statistical Analysis 2: Comparison: Test Dentifrice 2 (RDA~77) vs Reference Dentifrice 1 (RDA~80); Test type: Superiority; p = 0.0043, ANCOVA — Statistical significance set at 5% level; From ANCOVA with treatment and smoking status as factors and baseline pre-prophylaxis overall MLSI score as covariate; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.08 to -0.02] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Test Dentifrice 1 (RDA~58) vs Reference Dentifrice 2 (RDA~120); Test type: Superiority; p < .0001, ANCOVA — Statistical significance set at 5% level; From ANCOVA with treatment and smoking status as factors and baseline pre-prophylaxis overall MLSI score as covariate; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.12 to -0.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Test Dentifrice 2 (RDA~77) vs Reference Dentifrice 2 (RDA~120); Test type: Superiority; p < .0001, ANCOVA — Statistical significance set at 5% level; From ANCOVA with treatment and smoking status as factors and baseline pre-prophylaxis overall MLSI score as covariate; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.15 to -0.08] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Test Dentifrice 1 (RDA~58) vs Test Dentifrice 2 (RDA~77); Test type: Superiority; p = 0.0779, ANCOVA — Statistical significance set at 5% level; From ANCOVA with treatment and smoking status as factors and baseline pre-prophylaxis overall MLSI score as covariate; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.00 to 0.06] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Reference Dentifrice 1 (RDA~80) vs Reference Dentifrice 2 (RDA~120); Test type: Superiority; p = 0.0001, ANCOVA — Statistical significance set at 5% level; From ANCOVA with treatment and smoking status as factors and baseline pre-prophylaxis overall MLSI score as covariate; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [0.03 to 0.10] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Approximately 35 days (28+/- 2 days, maximum 30 days plus 5 days follow up after last use of study product.
Description: Safety population (N=220) included all participants who were randomized and received at least one dose of investigational product and was reported by treatment received.
Arm/Group | Test Dentifrice 1 (RDA~58) | Test Dentifrice 2 (RDA~77) | Reference Dentifrice 1 (RDA~80) | Reference Dentifrice 2 (RDA~120)
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55 | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55 | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 1/55 | 0/55 | 1/55 | 0/55
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Test Dentifrice 1 (RDA~58) (N=55) | Test Dentifrice 2 (RDA~77) (N=55) | Reference Dentifrice 1 (RDA~80) (N=55) | Reference Dentifrice 2 (RDA~120) (N=55)
BACK INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT03160703/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT03160703/SAP_001.pdf